CLINICAL TRIAL: NCT01156350
Title: Haplo-identical Hematopoietic Stem Cell Transplantation Following Reduced-intensity Conditioning in Children With Neuroblastoma
Acronym: Rice NK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0075
Record Dates: First submitted 2010-06-28; First posted 2010-07-02 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma - Haplo HSCT - Reduced Intensity Conditioning - immunotherapy NK
MeSH Terms: conditions — Neuroblastoma

INTERVENTIONS:
Drug: Busulfan - Fludarabine - TBI — This RICE NK protocol is a multicenter study of Haplo- HSCT using RIC with fludarabine (180 mg/m2), Busulfan IV (3,2 to 4,8 mg/kg/d), TBI 2 grays and CD3/CD19 graft depletion. A minimum of 8 106 CD34+ cells/kg were infused on day 0. No post grafting immunosuppression was applied if the graft contained < 2.5 x 104 CD3+ cells/kg

SUMMARY:
To date, no curative option exists for patients with relapsed or refractory stage IV neuroblastoma after previous autologous stem cell transplantation. Our preliminary results of RIC allo-HSCT (protocol RICE) indicate the feasability and low toxicity of allograft in heavily pre-treated children. Furthermore RIC SCT and immunomagnetic CD3/CD19 graft depletion may allow HHCT with lower toxicity and faster engraftment. CD3/CD19 depleted grafts not only contain CD34+ stem cells but also graft-facilitating cells, CD34- progenitors, dendritic and natural killer cells which may allow stable engraftment and participate to GvT effect.

After haploidentical stem cell transplantation anti tumour activity exerted by donor derived NK cells could be stimulated by NK cells injections. Those effects may help to reduce the relapse rate and to impove the outcome of those patients. The investigators prospectively evaluated engraftment and immune reconstitution.

DETAILED DESCRIPTION:
This RICE NK protocol is a multicenter study of Haplo- HSCT using RIC with fludarabine (180 mg/m2), Busulfan IV (3,2 to 4,8 mg/kg/d), TBI 2 grays and CD3/CD19 graft depletion. A minimum of 8 106 CD34+ cells/kg were infused on day 0. No post grafting immunosuppression was applied if the graft contained < 2.5 x 104 CD3+ cells/kg. At Day 30 and 60 post-graft we perform an donor CD56+ cells injection. The investigators develop this strategy in an European collaboration working on haploidentical stem cell transplantation for childhood refractory and metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* High Risk Neuroblastoma
* HLA haplo-identical family donor

Exclusion Criteria:

* patient with fast progressive neuroblastoma
* Lansky < 60%

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the feasibility of the CD3 / CD19 selected haplo identical hematopoietic stem cell transplant after conditioning with reduced intensity in children with neuroblastoma in failure of reference treatments | at one year

SECONDARY OUTCOMES:
Study of the overall survival Study of graft versus tumor effect at day + 100 | at day + 100

CONTACTS AND LOCATIONS:
Overall Officials: Catherine PAILLARD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France